CLINICAL TRIAL: NCT00761241
Title: A Phase II Protocol in Borderline Resectable Pancreatic Cancer Using Gemcitabine/Docetaxel Chemotherapy and An Oxaliplatin-Based Chemoradiation.
Brief Title: Borderline Resectable Pancreatic Cancer: Gemcitabine/Docetaxel and Oxaliplatin Based Chemo/RT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Vincent Picozzi, MD/Principal Investigator, Virginia Mason Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB07124; IST14087
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Pancreatic Cancer
Keywords: pancreas cancer; combined modality therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Fluorouracil; Oxaliplatin; Interferon-alpha; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemcitabine, Docetaxel, 5FU, Oxaliplatin — Gemcitabine: 1000 mg/m2 IV bolus days 1 and 8, repeated every 21 days x 8cycles Docetaxel: 40 mg/m2 IV bolus days 1 and 8, repeated every 21 days x 8 cycles Gemcitabine/docetaxel will be repeated (based upon initial response) Oxaliplatin: 40 mg/m2 IV on day 1 of each week of radiation 5-FU: 175 mg/m2 continuous infusion on days 1-18 and 29-46 of radiation
Biological: Alpha-interferon — Alpha-interferon: injected subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 29, 31, 33, 36, 38, 40, 43 and 46 during radiation therapy
Radiation: Abdominal/pelvic radiation therapy — 3-D conformal technique. The dose per fraction will be 180cGy, with a total dose of 5040 cGy in 28 fractions. Radiation therapy will be delivered on days 1-18 and days 29-46
Procedure: Pancreaticoduodenectomy — Surgery performed if subject is considered candidate by protocol definition.

SUMMARY:
This study is being conducted to find out what effects (good and bad) that a combination of treatment with chemotherapy, radiation therapy and surgery has on you and your pancreatic cancer. The chemotherapy drugs to be used: Gemcitabine, Docetaxel, Oxaliplatin, 5-FU and alpha-interferon. The goal is to decrease the size of the tumor, so that removal by surgery can be performed. Current treatments for this stage of pancreas cancer offer less than ideal results, with little opportunity for treatment with curative intent.

DETAILED DESCRIPTION:
Subjects must have biopsy proven adenocarcinoma of the pancreas which is bidimensionally measurable on CT. Cancer must be considered locally advanced (not able to be treated surgically). Subjects must not have received prior treatment for pancreatic cancer. Subjects must not have received prior radiation therapy to the abdomen or pelvis (for any reason). Subjects cannot be receiving immunosuppressive therapy (e.g. prednisone, methotrexate). Eligible subjects will receive initial chemotherapy regimen to include eight cycles of Gemcitabine and Docetaxel. All subjects will be re-evaluated for surgery - if tumor has shrunk enough, subject will undergo surgery, followed by additional chemotherapy of Oxaliplatin, 5FU and Alpha-interferon and radiation therapy; once subject has recovered from side effects of the chemo/radiation therapy, they will receive a final chemotherapy regimen of four cycles of Gemcitabine and docetaxel. Subjects who are not surgical candidates after eight cycles of chemotherapy will undergo an additional four cycles of Gemcitabine and docetaxel followed by reassessment for surgery. If they are a surgical candidate, they will undergo surgery followed by chemo/radiation therapy regimen. If they are not a surgical candidate, they will undergo the chemo/radiation therapy regimen.

Subjects may be removed from the study treatment for the following reasons:

* The investigator feels the subject is not benefitting from treatment
* The subject chooses to discontinue for any reason
* The subject experiences side effects which are considered to be unacceptable
* The subject has an increase in the size of their tumor

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the pancreas
* Tumor must be radiographically bidimensional by abdominal/pelvic CT
* Cancer must be locally advanced and not considered immediately treated by standard surgical procedure
* No prior therapy for pancreas cancer

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects who have received prior external beam radiation to the abdomen or pelvis
* Subjects receiving chronic immunosuppressive therapy (prednisone, methotrexate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Two year overall survival | two years

SECONDARY OUTCOMES:
median disease free survival initial response rate to gemcitabine/docetaxel (tumor marker and radiographic) toxicity of overall regimen time to disease progression percentage of patients able to complete protocol to entirety | two years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Picozzi, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States